Version number / Version date: The first version 1.0 / April  $15,\,2020$ 

**Plan ID: 2018LCYJ005** 

# **Informed Consent Form (ICF)**

| Protocol Title: Integrated image strategy of head and neck CTA combined with |
|------------------------------------------------------------------------------|
| multimodal MRI to assess the risk of cerebrovascular disease |
| Volunteer name: |
| Initials: |
| Serial number: |

#### Test purpose

A comprehensive imaging strategy using head and neck CTA combined with multimodal MRI to assess the risk of cerebrovascular disease was adopted using 3.0T MRI as the platform.

## **Test procedure**

The course of the experiment included lifestyle assessment, clinical relevant information acquisition/cognitive assessment, and multi-mode MRI scanning. During an MRI scan, you will be asked to keep your body, and especially your head, still for as long as possible. To help you stay still, some sponge filler will be placed between your head and the coil.

#### **Benefit**

There is no direct benefit to you from your participation in this trial.

Potential hazards and side effects

An MRI scan requires you to lie in a small, enclosed environment, and some people may feel uncomfortable, or scared, nervous, sweaty, or otherwise uncomfortable. If you have a metal implant in your body, such as a metal-containing denture, stent, contraceptive ring, etc., do not have an MRI. Please do not hide the metal implants in your body or you will suffer the consequences.

### **Privacy**

Your personal information and the data you provide during the study will not be disclosed without your written permission. The exceptions are: 1. Where it is possible to protect your interests (for example, if you are injured or in an emergency); 2. 2. Legal requirements. Your personally identifiable information will not be included when the results are published and discussed at meetings.

#### **Injured statement**

If you suffer an injury as a direct result of this study, you should contact the principal responsible person and you will receive the necessary medical treatment. However, this treatment does not suggest that it was the fault of the center or the person in charge that caused your injury. The Center or the person in charge will not provide other compensation.

### Participate in and terminate the test

Your participation in this trial is entirely voluntary, and if you choose not to participate, there will be no adverse effects on you. If you decide to participate, you may opt out at any time without any reason.

## The subjects

I declare that I have been informed of the purpose, process, possible risks and side effects, and potential benefits and costs of this trial. All my questions were satisfactorily answered. I have read the informed consent in detail. My signature below indicates my willingness to take part in the experiment.

| α' , | <b>D</b> 4 |
|------------|------------|
| Signature: | Date: |
| Signature. | Date. |